CLINICAL TRIAL: NCT01944241
Title: Cervical Surgery and the Fertility Effect
Brief Title: Cervical Surgery and the Fertility Effect (c-SAFE)
Acronym: c-SAFE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Merrion Fertility Clinic (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: MFC2
Record Dates: First submitted 2012-10-24; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Infertility
Keywords: cervical surgery; LLETZ; LEEP; Cone biopsy; Fertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with cervical surgery: The cases will include women who have had cervical surgery, either LLETZ or cone biopsy
- women with no surgery: controls will be women who have attended colposcopy but who have not had surgery.

SUMMARY:
Over the last 20 years, cervical screening programs have had huge success in reducing cervical cancer rates. These programs have done this by screening women at risk of developing cancer with regular smear tests. Women with abnormal smears are followed up in colposcopy clinics, and where needed, cervical surgery is performed to remove pre-cancerous areas on the cervix.

Surgery to the cervix can include LLETZ (Large loop excision of the transformation zone) treatment or cone biopsy. Many studies in the last few years have looked at the impact that this necessary surgery can have on the function of the cervix. These studies have mainly found an association between LLETZ treatment and an increased risk of preterm labour. There have been no large studies investigating the effect cervical surgery may have on fertility.

The investigators would like to examine the impact that cervical surgery may have on a woman's future fertility. It has been postulated that cervical surgery may cause the cervix to close, preventing sperm getting through or that it may cause changes in the secretions of the cervix, secretions that are necessary for normal interaction with sperm.

The investigators would like to send a questionnaire to women who have attended colposcopy. The investigators will ask these women a series of questions relating to fertility desires and divide the women in to two groups depending on whether the women needed cervical surgery for pre-cancerous lesions or not.

Hypothesis: That cervical surgery has an impact on the function of the cervix and on fertility.

DETAILED DESCRIPTION:
With an increasing amount of young women undergoing cervical surgery for the treatment of CIN, the fertility consequences need to be investigated. Infertility is estimated to affect approximately one in six to one in ten couples and only about half of these seek medical assistance. Causes of infertility include anovulation, tubal occlusion, endometriosis, cervical and male factor. In approximately one third of cases, there is no cause found as to why a couple are unable to conceive.

Many recent studies have looked at the likely association between cervical surgery and increased risk of preterm labour. It has also been suggested in an Australian study that even women with untreated CIN have a higher risk for preterm delivery, although it is unclear whether this is related to the CIN itself, HPV effect or inflammatory changes in the cervix. Studies are needed to clarify this further.

There are few studies published in the literature, investigating the possibility that cervical surgery has an effect on long term fertility. Most of these studies are small and under-powered.

Kennedy et al in 1993 raised the possibility of cervical stenosis and amucorrhoea following LLETZ in their retrospective study. In this study, 15 out of 2315 women who had LLETZ, were subsequently seen in a fertility clinic. 2 out of these 15 women studied had cervical stenosis. The authors advised caution with the use of LLETZ in young women with mild to moderate dyskaryosis, although the investigators did concede that their numbers were small to draw definite conclusions.

Bigrigg et al in 1994 performed a case controlled questionnaire regarding the safety and efficacy of LLETZ and this involved questions regarding infertility. There were 250 matched pairs- women who had had a LLETZ (study group) and those women identified who had normal cytology from their database (control group), for the entire study, but only 134 women answered the questions on infertility (72 in the LLETZ group and 62 in the control group). The investigators reported no apparent difference in infertility between the groups. Again this study was limited by size -72 in the study group and 62 in the control group could remember how long it took to conceive.

Cruickshank et al in 1995, followed up 653 women following LLETZ with a questionnaire and found that none of the women subsequently investigated for infertility were found to have cervical stenosis or amucorrhoea. Again this study was limited by size and incomplete response rates. Of the 653 women, the majority reported that they had not stopped contraception since their treatment - 452. Only 57 women reported trying to become pregnant, of whom 11 succeeded, but 144 women did not answer this question on intention to become pregnant. It is difficult to draw conclusions from this incomplete data and small numbers

As the cervix is necessary for sperm transit and subsequent fertility, it is likely that factors, which affect the cervix, would also affect fertility. Therefore, women who attend colposcopy for abnormal cervical cytology may be already at increased risk of fertility problems which treatments such as surgery may accentuate.

In relation to cervical surgery, three potential mechanisms of damage have been proposed:

1. Cervical stenosis - needs to be complete to prevent sperm entry.
2. Secondary infection leading to ascending infection and tubal damage.
3. Changes in physical characteristics of cervical mucus.

However it must be noted that not all surgery on the cervix is the same. Specimens from LLETZ and cone treatments vary in size considerably and as would be intuitively suspected but also has been confirmed by studies, the thickness and volume of the specimens can predict the relative risk of pregnancy related morbidity. No study has looked at whether this size effect also relates to fertility.

Some studies suggest that sub-fertile women who attend for IVF are more likely to have abnormal cervical cytology. As this is HPV related, they may also be more likely to have had other sexually transmitted infections. These may have caused tubal damage, thus leading to infertility problems.

The psychological impact of receiving abnormal smear results and having to attend colposcopy has also been investigated. Recent studies now show that women are concerned and have anxiety about the potential effect that such results and treatments will have on patients' long term fertility. To be able to adequately reassure women that there will be no negative consequences to their reproductive health it is vital that the investigators research the fertility effects as well as the obstetric effects that possible treatments may have.

The investigators would like to investigate the relationship between cervical surgery and infertility in a large group of women who have attended the colposcopy clinic in the National Maternity Hospital, Holles Street between the years 2001 and 2007.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40 years
* History of attendance at colposcopy in the specified years.

Exclusion Criteria:

* Not fitting inclusion criteria

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be a retrospective cohort study in women of reproductive age, who attended the colposcopy services in the National Maternity Hospital from the years 2001 to 2007. The cases will include women who have had cervical surgery, either LLETZ or cone biopsy and the controls will be women who have attended colposcopy but who have not had surgery.
  The cases will be identified by using the Mediscan database in the colposcopy clinic to identify those women who have had a LLETZ procedure and those who have had a cone biopsy will be identified by accessing pathology records for cone biopsies for the specified years. The controls will be selected by using Mediscan again, identifying women who have attended colposcopy but who have not had cervical surgery
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The number of women with subfertility after cervical surgery | 12 months
  This study will be a retrospective cohort study in women of reproductive age, who attended the colposcopy services in the National Maternity Hospital from the years 2001 to 2007. The cases will include women who have had cervical surgery, either LLETZ or cone biopsy and the controls will be women who have attended colposcopy but who have not had surgery.

SECONDARY OUTCOMES:
The number of women with subfertility correlatied with the size of the specimen removed. | 12 months
  To investigate whether the size of the amount of cervix removed correlates with subfertility problems.
The number of women with subfertility who have had either a cone or LLETZ biopsy. | 12 months
  To investigate the impact that type of surgery has on fertility
The number of women who have had repeat surgery and have subfertility. | 12 months
  The investigators wish to determine whether repeat cervical surgery has an impact on subfertility.

CONTACTS AND LOCATIONS:
Overall Officials: mary wingfield, MRCOG,MD, Principal Investigator — Merrion Fertility Clinic, National Maternity Hospital
Locations (1):
- Merrion Fertility Clinic & National Maternity Hospital, Dublin, Ireland